CLINICAL TRIAL: NCT02418936
Title: Development and Clinical Application of Two New Genetic Deafness Gene
Brief Title: Development and Clinical Application of Two New Genetic Deafness Gene Diagnostic Kit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2014L01
Record Dates: First submitted 2015-04-13; First posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Waardenburg Syndrome; Large Vestibular Aqueduct Syndrome
Keywords: Waardenburg syndrome; Large vestibular aqueduct syndrome; Diagnosis; copy number variation; Multiplex polymerase chain reaction
MeSH Terms: conditions — Waardenburg Syndrome; Disease

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- WS: WS diagositic kit
  Interventions: Device: gene diagnostic kit
- LVAS: LVAS diagositic kit
  Interventions: Device: gene diagnostic kit

INTERVENTIONS:
Device: gene diagnostic kit

SUMMARY:
The purpose of this study is to develop and applicate two new genetic deafness gene diagnostic kit for Waardenburg syndrome and large vestibular aquduct syndrome.

DETAILED DESCRIPTION:
1. For the pathogenic gene of Waardenburg syndrome and large vestibular aqueduct syndrome, based on the second-generation sequencing technology, the investigators develop multiplex PCR system for these two hereditary deafness gene diagnostic kit.
2. Using CNVplex high-throughput gene copy number detection technology to analyse Warrdenburg syndrome pathologic gene. CNVs analysis for Warrdenburg deafness syndrome develop special testing system / kit achieve SNP / CNVs detected simultaneously, as a supplementary means of genetic testing in clinical deafness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Waardenburg syndrome
* Clinical diagnosis of large vestibular aqueduct syndrome

Exclusion Criteria:

* Could not be able to exsanguinate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who are diagnosised Waardenburg syndrome or large vestibular aqueduct syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the positive rate of WS diagnosis | two years

SECONDARY OUTCOMES:
the positive rate of LVAS diagnosis | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China